CLINICAL TRIAL: NCT05453500
Title: Dose-Adjusted Etoposide, Prednisone, Vincristine, Cyclophosphamide, and Doxorubicin (DA-EPOCH) +/- Rituximab (R) + Tafasitamab-cxix for the Treatment of Newly-Diagnosed Adults With Philadelphia Chromosome-Negative (Ph-) B-cell Lymphoblastic Lymphoma/Leukemia (B-ALL)
Brief Title: Chemotherapy (DA-EPOCH+/-R) and Targeted Therapy (Tafasitamab) for the Treatment of Newly-Diagnosed Philadelphia Chromosome Negative B Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1122464; NCI-2022-05225 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11008 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: B Acute Lymphoblastic Leukemia, Philadelphia Chromosome Negative
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Cyclophosphamide; Doxorubicin; Etoposide; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; tafasitamab; Immunoglobulins; Disulfides; Vincristine; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (DA-EPOCH+/-R, tafasitamab) (Experimental): Patients receive etoposide, doxorubicin, and vincristine IV continuously over 96 hours on days 1-4 of each cycle, cyclophosphamide IV over 1 hour on day 5 of each cycle, prednisone PO BID on days 1-5 of each cycle, and tafasitamab IV weekly on days 1, 8, and 15 of each cycle. CD20 positive patients also receive rituximab IV per guidelines on days 1 or 5 of each cycle. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration or biopsy, CT scan, lumbar puncture and undergo blood sample and cerebrospinal fluid collection throughout the trial.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Drug: Prednisone; Biological: Rituximab; Biological: Tafasitamab; Drug: Vincristine; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Lumbar Puncture; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
Biological: Tafasitamab — Given IV
  Other Names: Immunoglobulin, Anti-(Human Cd19 Antigen) (Human-mus musculus Monoclonal MOR00208 Heavy Chain), Disulfide with Human-mus musculus Monoclonal MOR00208 .Kappa.-chain, Dimer; Monjuvi; MOR-00208; MOR00208; MOR208; Tafasitamab-cxix; XmAb5574
Drug: Vincristine — Given IV
  Other Names: Leurocristine; VCR; Vincrystine
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT Scan; CT Scan; computerized axial tomography
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; spinal tap
Procedure: Biospecimen Collection — Undergo blood sample and cerebrospinal fluid collection
  Other Names: Biological Sample Collection

SUMMARY:
This phase II clinical trial tests a chemotherapy regimen (dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide and doxorubicin with or without rituximab [DA-EPOCH+/-R]) with the addition of targeted therapy (tafasitamab) for the treatment of patients with newly diagnosed Philadelphia chromosome negative (Ph-) B acute lymphoblastic leukemia (B-ALL). Chemotherapy drugs, such as those in EPOCH+/-R, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Tafasitamab is in a class of medications called monoclonal antibodies. It works by helping the body to slow or stop the growth of cancer cells. Adding tafasitamab to the DA-EPOCH+/-R regimen may work better than DA-EPOCH+/-R alone in treating newly diagnosed Ph- B-ALL.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive etoposide, doxorubicin, and vincristine intravenously (IV) continuously over 96 hours on days 1-4 of each cycle, cyclophosphamide IV over 1 hour on day 5 of each cycle, prednisone orally (PO) twice daily (BID) on days 1-5 of each cycle, and tafasitamab IV weekly on days 1, 8, and 15 of each cycle. CD20 positive patients also receive rituximab IV per guidelines on days 1 or 5 of each cycle. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration or biopsy, computed tomography (CT) scan, lumbar puncture and undergo blood sample and cerebrospinal fluid collection throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years and every 6 months for 3 years (total follow-up time 5 years).

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years and older) with newly-diagnosed CD19+ Ph- B-ALL
* In the opinion of the treating investigator, patients must be an unsuitable candidate for a pediatric-inspired regimen, reasons for which may include (but not be limited to) older age (e.g., >= 40 years), practical/logistical barriers to or toxicity concerns from administration of a pediatric-inspired regimen
* Marrow or blood involvement detectable by MFC
* Total bilirubin =< 2.0 x upper limit of normal (ULN) (unless attributed to Gilbert's disease or other causes of inherited indirect hyperbilirubinemia, at which point total bilirubin must be =< 4.0 x ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5.0 x institutional ULN. (Note: Patients with liver test abnormalities attributable to hepatic involvement by ALL will be permitted if the total bilirubin is =< 5.0 x ULN and ALT/AST are =< 8.0 x ULN)
* Calculated creatinine clearance of > 30 ml/min, as measured by the Modification of Diet in Renal Disease (MDRD) equation, will be eligible
* As patients with ALL frequently have cytopenias, no hematologic parameters will be required for enrollment or to receive the first cycle of treatment. However, adequate recovery of blood counts will be required to receive subsequent cycles
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2. (Performance status of 3 will be allowed if poor performance status is thought to be directly secondary to ALL)
* Ability to give informed consent and comply with the protocol
* Anticipated survival of at least 3 months, independent of ALL

Exclusion Criteria:

* Burkitt lymphoma/leukemia
* No prior systemic therapy for ALL except to control acute symptoms and/or hyperleukocytosis (e.g., corticosteroids, cytarabine, etc.)
* No isolated extramedullary or known parenchymal central nervous system (CNS) disease
* Known hypersensitivity or intolerance to any of the agents under investigation
* Other medical or psychiatric conditions that in the opinion of the investigator would preclude safe participation in the protocol
* May not be pregnant or nursing

  * Pregnancy test is only required in women, unless they are highly unlikely to conceive (defined as [1] surgically sterilized, or [2] postmenopausal [i.e., a woman who is > 50 years old or who has not had menses for >=1 year], or [3] not heterosexually active)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of minimal residual disease (MRD) | After 1 cycle of treatment (each cycle = 21 days)
  Efficacy of the addition of tafasitamab (tafa) to dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin with our without rituximab (DA-EPOCH±R) will be assessed using the rate of minimal residual disease (MRD) as measured by multiparameter flow cytometry (MFC) in the University of Washington hematopathology lab. Will consider an absolute increase in the rate of MRD- after one cycle to 50% to be a signal of interest (i.e., increase from 28%).

SECONDARY OUTCOMES:
Rate of MRD | After 4 cycles of treatment (each cycle = 21 days)
  Measured by MFC. Will be assessed only descriptively, using means and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures, and either Kaplan-Meier or cumulative incidence estimates for time-to-event outcomes (depending on whether competing risks are present).
Incidence of adverse events | Up to 5 years
  Safety measured by the incidence of non-hematologic toxicities >= grade 3 evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v) 5.0. Will be assessed only descriptively, using means and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures, and either Kaplan-Meier or cumulative incidence estimates for time-to-event outcomes (depending on whether competing risks are present).
Event-free survival (EFS) | Up to 5 years
  Will be assessed only descriptively, using means and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures, and either Kaplan-Meier or cumulative incidence estimates for time-to-event outcomes (depending on whether competing risks are present).
Relapse-free survival (RFS) | Up to 5 years
  Will be assessed only descriptively, using means and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures, and either Kaplan-Meier or cumulative incidence estimates for time-to-event outcomes (depending on whether competing risks are present).
Overall survival (OS) | Up to 5 years
  Will be assessed only descriptively, using means and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures, and either Kaplan-Meier or cumulative incidence estimates for time-to-event outcomes (depending on whether competing risks are present).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan D. Cassaday, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No